CLINICAL TRIAL: NCT00622505
Title: Bone Marker-directed Dosing of ZOMETA® (Zoledronic Acid) for the Prevention of Skeletal Complications in Patients With Advanced Multiple Myeloma.
Brief Title: Zoledronic Acid Treatment (Every 4 or 12 Weeks) to Prevent Skeletal Complications in Advanced Multiple Myeloma Participants
Acronym: Z-MARK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CZOL446EUS129
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Results first posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; zoledronic acid; skeletal complications; bone
MeSH Terms: conditions — Multiple Myeloma | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zoledronic acid (Experimental): Participants received 4 milligrams (mg) or a reduced dose, i.e., 3.5 mg, or 3.3 mg or 3.0 mg of Zoledronic acid as an IV infusion over a minimum of 15 minutes, every 4 weeks or every 12 weeks for up to 96 weeks based on the participants most recent urine N-telopeptide of type 1 collagen (NTx) measurement (greater than or equal to [≥] 50 nanomoles per millimoles [nmol/mmol] creatinine or <50 nmol/mmol creatinine, respectively).
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: zoledronic acid — Zoledronic acid concentrate (4 mg/5 milliliters [ml]) was diluted in 100 mL sterile 0.9% calcium-free sodium chloride or 5% dextrose injection, administered IV, either 4 or 12 weeks for 96 weeks.
  Other Names: Zometa

SUMMARY:
This study evaluated the effectiveness and safety of a dosing method for zoledronic acid in preventing skeletal complications in multiple myeloma participants who have been on an intravenous (IV) bisphosphonate for about one to two years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma
* Have been on zoledronic acid or pamidronate for 1-2 years and therapy must have been initiated for osteolytic lesion, bone fracture, spinal compression, or osteopenia due to multiple myeloma
* Stable renal function

Exclusion Criteria:

* Known sensitivity to bisphosphonates
* Receiving investigational drugs considered not safe for co-administration or have a significant effect on bone turnover
* Current active dental problems
* Had bone marrow transplant or blood stem cell transplant within 2 months before study entry or planned transplant within 2 months following enrollment

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2007-11-07 (Actual); Primary Completion 2012-04-03 (Actual); Study Completion 2012-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (42):
- United States (42):
  - TriValley Cancer Research and Treatment Center, Casa Grande, Arizona
  - Wilshire Oncology Medical Group, La Verne, California
  - Cedars Sinai Medical Center Outpatient Cancer Ctr. (4), Los Angeles, California
  - Palo Alto Medical Foundation Hematology/Oncology, Mountain View, California
  - Oncology Care Medical Associates, San Gabriel, California
  - Santa Clara Valley Health & Hospital System, San Jose, California
  - University of Colorado U of Colorado Cancer Center, Aurora, Colorado
  - Hematology Oncology PC, Stamford, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Palm Beach Institute of Hematology Oncology, Boynton Beach, Florida
  - Innovative Medical Research of South Florida Innovative Med Research, Miami Shores, Florida
  - Cancer Centers of Florida PA Cancer Centers of Central FL, Ocoee, Florida
  - Integrated Community Oncology Network Florida Oncology Associates, Orange Park, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Loyola University Medical Center /Cardinal Bernardin Cancer Loyola Univ Med Ctr, Maywood, Illinois
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Center for Cancer & Blood Disorders, Bethesda, Maryland
  - Oncology - Hematology Associates, PA Oncology Hematology Assoc, Clinton, Maryland
  - Dana Farber Cancer Institute Clinical Research Coordinator, Boston, Massachusetts
  - Boston VA Healthcare Boston VA, Boston, Massachusetts
  - Berkshire Hematology Oncology, Pittsfield, Massachusetts
  - N MS Hematology & Oncology, Tupelo, Mississippi
  - Hematology & Oncology Consultants, PC Hematology & Oncology, Omaha, Nebraska
  - Somerset Hematology Oncology Associates Somerset Hema Oncol Assoc (2), Somerset, New Jersey
  - Cooper Cancer Center, Voorhees Township, New Jersey
  - Rochester General Hospital / Lipson Cancer Center Lipson Cancer Center, Rochester, New York
  - University of Rochester MC / James P. Wilmot Cancer Center James P. Wilmot Cancer Center, Rochester, New York
  - SUNY - Upstate Medical University Div. of Hematology-Oncology, Syracuse, New York
  - Carolina Oncology Specialists, PC, Hickory, North Carolina
  - Regional Hematology-Oncology Associates PC, Langhorne, Pennsylvania
  - Temple University Temple University, Philadelphia, Pennsylvania
  - Medical Associates, PA, Charleston, South Carolina
  - Low Country Hematology Oncology Dept of Lowcountry Hem/Onc, Mt. Pleasant, South Carolina
  - Lexington Oncology Associates, West Columbia, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - Blood and Cancer Center of East Texas, Tyler, Texas
  - East Texas Medical Center Cancer Institute, Tyler, Texas
  - Northern Utah Cancer Associates Dept.ofNorthernUtahAssoc., Ogden, Utah
  - Central Utah Clinic Central Utah Clinic (8), Provo, Utah
  - Peninsula Cancer Institute, Newport News, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - West Virginia University Health Research Center Clinical Trial Research Unit, Morgantown, West Virginia

REFERENCES:
- [Result] Raje N, Vescio R, Montgomery CW, Badros A, Munshi N, Orlowski R, Hadala JT, Warsi G, Argonza-Aviles E, Ericson SG, Anderson KC. Bone Marker-Directed Dosing of Zoledronic Acid for the Prevention of Skeletal Complications in Patients with Multiple Myeloma: Results of the Z-MARK Study. Clin Cancer Res. 2016 Mar 15;22(6):1378-84. doi: 10.1158/1078-0432.CCR-15-1864. Epub 2015 Dec 7. PMID 26644410

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 67 centers in the United States (US) from 07 November 2007 to 03 April 2012.
Pre-assignment Details: A total of 121 participants with Advanced Multiple Myeloma were enrolled in this study. By study design, any participants who had a Skeletal-related Event (SRE) in Zoledronic Acid Every 12 Weeks group was switched to Zoledronic Acid Every 4 Weeks or 12 Weeks group and reported as Zoledronic Acid Every 4 Weeks or 12 Weeks group, respectively.
Groups:
- Zoledronic Acid Every 12 Weeks: Participants received 4 mg or a reduced dose, i.e., 3.5 mg, or 3.3 mg or 3.0 mg of Zoledronic acid as an IV infusion over a minimum of 15 minutes every 12 weeks for up to 96 weeks based on the participants most recent urine NTx measurement ( <50 nmol/mmol creatinine).
- Zoledronic Acid Every 4 Weeks or 12 Weeks: Participants received 4 mg or a reduced dose, i.e., 3.5 mg, or 3.3 mg or 3.0 mg of Zoledronic acid as an IV infusion over a minimum of 15 minutes every 4 weeks or every 12 weeks for up to 96 weeks based on the participants most recent urine NTx measurement (≥ 50 nmol/mmol creatinine or <50 nmol/mmol creatinine, respectively).
Period: Overall Study
Arm/Group | Zoledronic Acid Every 12 Weeks | Zoledronic Acid Every 4 Weeks or 12 Weeks
Started | 79 | 42
Completed | 50 | 19
Not Completed | 29 | 23
Not completed — Adverse Event | 9 | 7
Not completed — Abnormal Laboratory Value(s) | 3 | 5
Not completed — Abnormal Test Procedure Result(s) | 1 | 0
Not completed — Withdrawal by Subject | 12 | 5
Not completed — Administrative Problems | 2 | 4
Not completed — Death | 2 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all participants who were enrolled in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid Every 12 Weeks | Zoledronic Acid Every 4 Weeks or 12 Weeks | Total
Number analyzed (Participants) | 79 | 42 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.91) | 65.8 (12.66) | 63.8 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 21 | 57
  Male | 43 | 21 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥1 SRE at the End of 1 Year on Study
Description: SRE was defined as pathological bone fracture, initiation of radiotherapy or surgery on bone, spinal cord compression, or hypercalcemia of malignancy (HCM). SRE was assessed by centrally read radiographic bone surveys.
Time Frame: 1 year
Population: ITT analysis set included all participants who were enrolled in this study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zoledronic Acid Every 12 Weeks | Zoledronic Acid Every 4 Weeks or 12 Weeks
Number analyzed (Participants) | 79 | 42
percentage of participants | 0 [NA to NA] — Upper and lower limits of 95% CI were not estimable due to the smaller number of participants with the event. | 0.17 [0.05 to 0.28]

2. Secondary Outcome: Time to First SRE on Study
Description: The time to first SRE is defined as the date of enrollment to the date of the first occurrence of any SRE on the study. SRE includes pathological fracture, initiation of radiotherapy or surgery on bone, spinal cord compression, or HCM. Participants who drop-out was treated as censored observations. Time to first SRE on the study was assessed by the Kaplan-Meier method.
Time Frame: Up to 2 years
Population: ITT analysis set included all participants who were enrolled in this study.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Zoledronic Acid Every 12 Weeks | Zoledronic Acid Every 4 Weeks or 12 Weeks
Number analyzed (Participants) | 79 | 42
years | NA [NA to NA] — The median and 95 % CI was not estimable because there were too few events (low incidence of observed SREs) to calculate the median and 95 % CI. | NA [NA to NA] — The median and 95 % CI was not estimable because there were too few events (low incidence of observed SREs) to calculate the median and 95 % CI.

3. Secondary Outcome: Percentage of Participants Who Experienced Pathologic Bone Fracture
Description: Pathologic bone fractures are defined as bone fractures that occur spontaneously or as a result of trivial trauma.
Time Frame: Years 1 and 2
Population: ITT analysis set included all participants who were enrolled in the study. Number analyzed signifies the number of participants with data available for analysis at given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zoledronic Acid Every 12 Weeks | Zoledronic Acid Every 4 Weeks or 12 Weeks
Number analyzed (Participants) | 79 | 42
percentage of participants
  Year 1 | 0.00 [NA to NA] — Upper and lower limits of 95% CI were not estimable due to smaller number of participants with the event. | 0.07 [0.00 to 0.15]
  Year 2: number analyzed (Participants) | 63 | 38
  Year 2 | 0.00 [NA to NA] — Upper and lower limits of 95% CI were not estimable due to smaller number of participants with the event. | 0.03 [0.00 to 0.08]

4. Secondary Outcome: Percentage of Participants Who Experienced Spinal Cord Compression
Description: Spinal cord compression is caused by the impingement of a tumor on the spinal cord and is associated with neurologic impairment and/or back pain.
Time Frame: Years 1 and 2
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zoledronic Acid Every 12 Weeks | Zoledronic Acid Every 4 Weeks or 12 Weeks
Number analyzed (Participants) | 79 | 42
percentage of participants
  Year 1 | 0.00 [NA to NA] — Upper and lower limits of 95% CI was not estimable due to smaller number of participants with the event. | 0.07 [0.00 to 0.15]
  Year 2: number analyzed (Participants) | 63 | 38
  Year 2 | 0.00 [NA to NA] — Upper and lower limits of 95% CI was not estimable due to smaller number of participants with the event. | 0.00 [NA to NA] — Upper and lower limits of 95% CI was not estimable due to smaller number of participants with the event.

5. Secondary Outcome: Percentage of Participants Who Experienced Radiation to Bone
Description: Radiation therapy to bone events includes irradiation of bone to palliate painful lesions, to treat or prevent pathologic fractures, or to treat or prevent spinal cord compression.
Time Frame: Years 1 and 2
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zoledronic Acid Every 12 Weeks | Zoledronic Acid Every 4 Weeks or 12 Weeks
Number analyzed (Participants) | 79 | 42
percentage of participants
  Year 1 | 0.00 [NA to NA] — Upper and lower limits of 95% CI were not estimable due to smaller number of participants with the event. | 0.10 [0.01 to 0.18]
  Year 2: number analyzed (Participants) | 63 | 38
  Year 2 | 0.00 [NA to NA] — Upper and lower limits of 95% CI were not estimable due to smaller number of participants with the event. | 0.11 [0.01 to 0.20]

6. Secondary Outcome: Percentage of Participants Who Experienced Surgery to Bone
Description: Surgery to bone events includes surgical procedures that are performed to set or stabilize pathologic fractures or areas of spinal cord compression and surgical procedures that are performed to prevent an imminent pathologic fracture or spinal cord compression.
Time Frame: Years 1 and 2
Population: ITT analysis set includes all participants who were enrolled in this study. Number analyzed signifies the number of participants with data available for analysis at given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zoledronic Acid Every 12 Weeks | Zoledronic Acid Every 4 Weeks or 12 Weeks
Number analyzed (Participants) | 79 | 42
percentage of participants
  Year 1 | 0.00 [NA to NA] — Upper and lower limits of 95% CI was not estimable due to smaller number of participants with the event. | 0.02 [0.00 to 0.07]
  Year 2: number analyzed (Participants) | 63 | 38
  Year 2 | 0.00 [NA to NA] — Upper and lower limits of 95% CI was not estimable due to smaller number of participants with the event. | 0.00 [NA to NA] — Upper and lower limits of 95% CI was not estimable due to smaller number of participants with the event.

7. Secondary Outcome: Percentage of Participants Who Experienced HCM
Description: HCM is defined as corrected serum calcium ≥ 12.0 milligrams per deciliter (mg/dL) (3.00 millimoles per liter [mmol/L]), or a lower level of hypercalcemia that was symptomatic and required active treatment other than rehydration.
Time Frame: Years 1 and 2
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zoledronic Acid Every 12 Weeks | Zoledronic Acid Every 4 Weeks or 12 Weeks
Number analyzed (Participants) | 79 | 42
percentage of participants
  Year 1 | 0.00 [NA to NA] — Upper and lower limits of 95% CI was not estimable due to smaller number of participants with the event. | 0.02 [0.00 to 0.07]
  Year 2: number analyzed (Participants) | 63 | 38
  Year 2 | 0.00 [NA to NA] — Upper and lower limits of 95% CI was not estimable due to smaller number of participants with the event. | 0.00 [NA to NA] — Upper and lower limits of 95% CI was not estimable due to smaller number of participants with the event.

8. Secondary Outcome: Skeletal Related Event (SRE) Rate
Description: The SRE rate for each participant was calculated as the number of SREs/total follow-up time. SRE included pathological bone fracture, initiation of radiotherapy or surgery on bone, spinal cord compression, or HCM.
Time Frame: Years 1 and 2
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: number of SRE/total follow-up time
Arm/Group | Zoledronic Acid Every 12 Weeks | Zoledronic Acid Every 4 Weeks or 12 Weeks
Number analyzed (Participants) | 79 | 42
number of SRE/total follow-up time
  Year 1 | 0.00 (0.00) | 0.03 (0.080)
  Year 2: number analyzed (Participants) | 63 | 38
  Year 2 | 0.00 (0.00) | 0.02 (0.049)

9. Secondary Outcome: Change From Baseline in Urinary N-telopeptide of Type 1 Collagen (uNTx)
Description: uNTx is a biomarker used to measure the rate of bone turnover found in urine.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 60, 72, 84 and 100/End of Study (EOS)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of zoledronic acid. Number analyzed signifies the number of participants with data available for analysis at given time point.
Measure: Mean (Standard Deviation); unit: nmol/mmol creatinine
Arm/Group | Zoledronic Acid Every 12 Weeks | Zoledronic Acid Every 4 Weeks or 12 Weeks
Number analyzed (Participants) | 79 | 42
nmol/mmol creatinine
  Baseline | 19.8 (8.82) | 24.1 (15.63)
  Change from Baseline to Week 12: number analyzed (Participants) | 74 | 41
  Change from Baseline to Week 12 | 0.2 (11.50) | 4.3 (19.47)
  Change from Baseline to Week 24: number analyzed (Participants) | 73 | 40
  Change from Baseline to Week 24 | -1.4 (8.72) | -0.5 (15.66)
  Change from Baseline to Week 36: number analyzed (Participants) | 65 | 40
  Change from Baseline to Week 36 | -2.0 (9.77) | -0.9 (13.92)
  Change from Baseline to Week 48: number analyzed (Participants) | 63 | 37
  Change from Baseline to Week 48 | -2.3 (9.24) | 1.7 (18.39)
  Change from Baseline to Week 60: number analyzed (Participants) | 59 | 32
  Change from Baseline to Week 60 | -2.5 (12.30) | -0.8 (17.54)
  Change from Baseline to Week 72: number analyzed (Participants) | 57 | 29
  Change from Baseline to Week 72 | -3.5 (10.99) | -6.7 (15.50)
  Change from Baseline to Week 84: number analyzed (Participants) | 55 | 23
  Change from Baseline to Week 84 | -3.0 (10.73) | -7.6 (18.51)
  Change from Baseline to Week 100: number analyzed (Participants) | 59 | 25
  Change from Baseline to Week 100 | -5.2 (9.25) | -7.4 (17.68)

10. Secondary Outcome: Time to Death
Description: Time to death was defined as the time from the date of enrollment to the date of death. Participants who dropped out or completed the study were considered censored observations. Time to death was assessed by Kaplan-Meier method.
Time Frame: Up to 2 years
Population: ITT analysis set included all participants who were enrolled in this study.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Zoledronic Acid Every 12 Weeks | Zoledronic Acid Every 4 Weeks or 12 Weeks
Number analyzed (Participants) | 79 | 42
years | NA [NA to NA] — The median and 95% CI was not estimable because there were too few events (low incidence of observed deaths) to calculate the median and 95% CI. | NA [NA to NA] — The median and 95% CI was not estimable because there were too few events (low incidence of observed deaths) to calculate the median and 95% CI.

ADVERSE EVENTS:
Time Frame: Up to 2 Years
Description: Safety analysis set included all enrolled participants who received at least 1 dose of zoledronic acid. Number analyzed signifies the number of participants with data available for analysis at given time point.
Arm/Group | Zoledronic Acid Every 12 Weeks | Zoledronic Acid Every 4 Weeks or 12 Weeks
All-Cause Mortality (participants affected / at risk) | 2/79 | 2/42
Serious Adverse Events (participants affected / at risk) | 23/79 | 25/42
Other Adverse Events (participants affected / at risk) | 70/79 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid Every 12 Weeks (N=79) | Zoledronic Acid Every 4 Weeks or 12 Weeks (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 3
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Ventricular asystole (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 2
Chest pain (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 3
Acute sinusitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 6
Pyelonephritis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Leukaemia plasmacytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 2
Spinal cord compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 4
Renal failure acute (Renal and urinary disorders) | 1 | 4
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 0 | 1
Venous insufficiency (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid Every 12 Weeks (N=79) | Zoledronic Acid Every 4 Weeks or 12 Weeks (N=42)
Anaemia (Blood and lymphatic system disorders) | 6 | 10
Leukopenia (Blood and lymphatic system disorders) | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 4 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 9
Tachycardia (Cardiac disorders) | 1 | 5
Abdominal discomfort (Gastrointestinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 9 | 11
Diarrhoea (Gastrointestinal disorders) | 15 | 11
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 5
Nausea (Gastrointestinal disorders) | 9 | 12
Toothache (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 5 | 3
Asthenia (General disorders) | 8 | 4
Chest discomfort (General disorders) | 2 | 4
Chest pain (General disorders) | 3 | 5
Fatigue (General disorders) | 15 | 16
Influenza like illness (General disorders) | 4 | 0
Oedema peripheral (General disorders) | 6 | 7
Pyrexia (General disorders) | 10 | 9
Bronchitis (Infections and infestations) | 6 | 7
Herpes zoster (Infections and infestations) | 8 | 5
Nasopharyngitis (Infections and infestations) | 6 | 5
Pneumonia (Infections and infestations) | 8 | 7
Sinusitis (Infections and infestations) | 6 | 6
Tooth infection (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 18 | 11
Urinary tract infection (Infections and infestations) | 8 | 5
Blood creatinine increased (Investigations) | 7 | 4
Weight decreased (Investigations) | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 10
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 9
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 3
Dizziness (Nervous system disorders) | 5 | 8
Headache (Nervous system disorders) | 7 | 3
Hypoaesthesia (Nervous system disorders) | 5 | 3
Neuropathy peripheral (Nervous system disorders) | 4 | 6
Anxiety (Psychiatric disorders) | 6 | 2
Depression (Psychiatric disorders) | 4 | 4
Insomnia (Psychiatric disorders) | 5 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 6 | 5
Hot flush (Vascular disorders) | 4 | 0
Hypertension (Vascular disorders) | 6 | 1
Hypotension (Vascular disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.